CLINICAL TRIAL: NCT06294795
Title: A Prospective Randomized Controlled Trial of Toric Intraocular Lens Implantation in Pediatric Cataractous Eyes
Brief Title: Toric Intraocular Lens Implantation in Pediatric Cataract
Acronym: TILIPC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kazakh Eye Research Institute (Network)
Responsible Party: Principal Investigator, Kairat Ruslanuly, a researcher, a vitreoretinal surgeon, Kazakh Eye Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-2024
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cataract Congenital; Astigmatism; IOL
Keywords: Cataract Congenital; Astigmatism; Toric IOL
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toric (Experimental): A folding hydrophobic acrylic IOLs AcrySof IQ Toric SN6ATx and Clareon Toric CNW0Tx
  Interventions: Procedure: congenital/pediatric cataract surgery; Device: Toric IOLs
- Non-toric (Active Comparator): A folding hydrophobic acrylic intraocular lens (IOL) AcrySof IQ SN60WF and Clareon SY60WF
  Interventions: Procedure: congenital/pediatric cataract surgery; Device: Non-Toric IOLs

INTERVENTIONS:
Procedure: congenital/pediatric cataract surgery — All procedures are performed under general anesthesia according to the standard technique of congenital/pediatric cataract surgery with an intraocular lens (IOL) implantation. Paracentesis is performed at 2.30 o'clock using a 20-gauge straight microvitreoretinal (MVR) knife; a high molecular weight ophthalmic viscosurgical devices (OVD) is injected into the anterior chamber. Then a 2.4 mm corneal tunnel incision is made at 11 o'clock with a disposable keratome knife 2.2 mm. Circular continuous capsulorhexis (≈ 5.5 mm). Сortical cleaving hydrodissection is followed by bimanual phacoaspiration in irrigation-aspiration mode. OVD is injected in the anterior chamber and an IOL is implanted in the capsular bag. Residual OVD is aspirated from the anterior chamber and behind the IOL and followed by IOL alignment. The surgery is completed with corneal hydration at the tunnel incision site.
  Other Names: phacoaspiration
Device: Non-Toric IOLs — A folding hydrophobic acrylic IOLs AcrySof IQ SN60WF and Clareon SY60WF for the non-toric group (Alcon Laboratories, Inc.) ARE implanted.
  Other Names: Models SN60WF and SY60WF
  Arms: Non-toric
Device: Toric IOLs — A folding hydrophobic acrylic IOLs AcrySof IQ Toric SN6ATx and Clareon Toric CNW0Tx for the toric group (Alcon Laboratories, Inc.) were implanted.
  Other Names: Models CNW0T3, CNW0T4, CNW0T5, CNW0T6, CNW0T7, CNW0T8 and SN6AT3, SN6AT4, SN6AT5, SN6AT6, SN6AT7, SN6AT8
  Arms: Toric

SUMMARY:
To evaluate the visual and refractive outcomes after an intraocular lens (IOL) implantation in pediatric eyes with cataract and preexisting corneal astigmatism

DETAILED DESCRIPTION:
This single-center, single-blinded, prospective, randomized controlled trial was performed at two sites of Kazakh Eye Research Institute.

Children with pediatric cataract and corneal astigmatism were included and randomized to two groups for pediatric cataract surgery with toric and non-toric intraocular lens (IOL) implantation. The uncorrected and corrected distance visual acuity, near visual acuity, keratometry data, and residual astigmatism were evaluated.

The purpose of this study is to evaluate the visual and refractive outcomes after a toric IOL implantation in pediatric eyes with cataract and preexisting corneal astigmatism.

ELIGIBILITY:
Inclusion criteria:

1. Visually significant cataract;
2. Corneal astigmatism more than 1.25 diopters;
3. Children aged ≥ 6 years and < 18 years.

Exclusion criteria:

1. Patients with a corneal diameter less than 9 mm;
2. Presence of corneal scarring;
3. Irregular astigmatism;
4. Intraocular pressure more than 25 mm Hg;
5. Active inflammatory process of the eyeball or signs of a previous episode of inflammation;
6. Traumatic, subluxated, or complicated cataract;
7. Persistent Fetal Vasculature;
8. Diseases of the optic nerve or macula that may limit visual potential;
9. History of previous intraocular surgeries;
10. Performing posterior capsulorhexis intraoperatively.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Uncorrected (UCDVA) and corrected (CDVA) distance visual acuity | recorded at each follow-up (on the fifth day, first month, third month, sixth month, and first year)
  measured using the Lea symbol visual acuity chart or the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart according to the patient's age
Uncorrected (UCNVA) and corrected (CNVA) near visual acuity | recorded at each follow-up (on the fifth day, first month, third month, sixth month, and first year)
  measured using the Lea symbol visual acuity chart or the ETDRS chart for near according to the patient's age
Refraction measurements | recorded at each follow-up (on the fifth day, first month, third month, sixth month, and first year)
  obtained with KR-1W Wavefront Analyzer

SECONDARY OUTCOMES:
Keratometry measurements | recorded at each follow-up (on the fifth day, first month, third month, sixth month, and first year)
  obtained with KR-1W Wavefront Analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Kairat Ruslanuly, MD, Principal Investigator — Kazakh Eye Research Institute
Locations (2):
- Kazakhstan (2):
  - Kazakh Eye Research Institute, Almaty
  - Kazakh Eye Research Institute, Astana

IPD SHARING:
Plan to Share IPD: Undecided